CLINICAL TRIAL: NCT04818697
Title: Effect of Social Isolation on Physical Activity Level, Health Literacy and Kinesophobia in Heart Rhythm Disorders During the COVID-19 Pandemic
Brief Title: Effect of Social Isolation on Physical Activity Level, and Kinesophobia in Heart Rhythm Disorders During Pandemic
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dilara Saklica, Principal Investigator, Hacettepe University
Other Study IDs: GO 20/633
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Heart Rhythm Disorder; Covid19; Social Isolation
Keywords: Heart Rhythm Disorder; Physical Activity; Kinesophobia; Health Literacy
MeSH Terms: conditions — COVID-19; Social Isolation; Motor Activity; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with heart rhythm disorders: Having been diagnosed with heart rhythm disorders such as atrial fibrillation, atrial tachycardia, ventricular tachycardia, and ventricular extrasystole
- Healthy individuals: Healthy individuals without chronic disease

SUMMARY:
The aim of our study is to examine the effect of social isolation on physical activity level, health literacy and kinesophobia in heart rhythm disorders.

DETAILED DESCRIPTION:
To prevent the spread of COVID-19, states are imposing quarantine measures and sanctions for all citizens to stay at home as much as possible. These measures severely limit physical activity. It is known that physical activity is an important preventive approach for many preventable diseases, especially cardiovascular diseases. Restriction of physical activity, loss of usual routine, and reduced social and physical contact with others can cause feelings of distress, disappointment, and isolation.

In the latest guidelines, increasing physical activity is recommended to prevent heart rhythm disorders and contribute to the effectiveness of treatment.

The aim of our study is to examine the effect of social isolation on physical activity level, health literacy, and kinesophobia in heart rhythm disorders.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with heart rhythm disorders
* Being clinically stable
* To comply with social isolation rules
* Volunteering to participate in the research

Exclusion Criteria:

* Having a cognitive problem
* Not being literate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthy individuals 18 years old and older, who are diagnosed with heart rhythm disorders, and whose local language is Turkish will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | June 2020-March 2021
  Physical activity level will be evaluated using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). The questionnaire provides information about the time spent on walking and moderate-to-severe / vigorous activities, while also evaluating the time spent sitting (sedentary behavior level). Physical activity levels are classified according to MET-min/week values. According to these values, people are classified as physically inactive (inactive), low level of physical activity (minimally active), and sufficient level of physical activity (very active).
Fear of Movement | June 2020-March 2021
  Fear of movement will be evaluated using the Tampa Scale of Kinesiophobia for Heart. The scale consists of 17 items. The score a participant can get is between 17 and 68. The higher the total score, the higher the severity of kinesiophobia.

SECONDARY OUTCOMES:
Health Literacy | June 2020-March 2021
  Health literacy will be evaluated using the Health Literacy Scale. This questionnaire consists of 25 questions and four sub-dimensions. A minimum of 25 and a maximum of 125 points are obtained for the entire scale. The higher the score obtained from the questionnaire, the higher the health literacy level of the participant.
Weekly Average of Steps | June 2020-March 2021
  The number of steps in the last week will be recorded and averaged using the pedometer applications from the participants own smartphones.
Weekly Average of Going Outside | June 2020-March 2021
  The number of days spent outside last week will be recorded.
The Comorbid Conditions | June 2020-March 2021
  The comorbid conditions of the patients will be evaluated by Charlson's comorbidity index. As the score obtained from the index increases, the comorbid situation increases.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Hikmet Yorgun, PhD MD, Study Chair — Hacettepe University; Ahmet Hakan Ates, PhD MD, Study Chair — Hacettepe University; Dilara Saklıca, MsC, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)